CLINICAL TRIAL: NCT03740477
Title: Screening for Atrial Fibrillation in Native AmeRicans Using iPhone ECG (SAFARI)
Brief Title: Screening for Atrial Fibrillation in Native AmeRicans Using iPhone ECG
Acronym: SAFARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9501
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrevention (Experimental): Eligible participants will receive a 30-second smartphone-based ECG
  Interventions: Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: ECG — Eligible participants will receive a 30-second ECG recording during their visit at the Absentee Shawnee Tribal clinic

SUMMARY:
Atrial fibrillation (AF) is the most common clinically significant arrhythmia and is associated with increased rates of stroke, heart failure, mortality, hospitalization, and cognitive decline. Approximately one third of ischemic strokes are attributable to either previously known or newly detected AF at the time of stroke. Many AF episodes are asymptomatic and stroke is the first manifestation of AF in at least 25% of AF-related strokes. Anticoagulation for AF leads to a reduction in stroke to levels similar to matched individuals without AF. Therefore, identifying AF in an earlier asymptomatic state (i.e. screening for silent AF), with subsequent initiation of anticoagulation in at-risk individuals, may decrease the risk of future thromboembolic events. The availability of inexpensive smartphone-based or handheld ECG devices that rapidly acquire a cardiac rhythm strip of quality comparable to a traditional 12-lead ECG have markedly enhanced the feasibility of AF screening. Native Americans have a high prevalence of diabetes and higher incidence of stroke than whites and blacks. Our central hypothesis is that screening for AF using a single time point, 30-second iPhone-based ECG recording over 2 weeks will result in identification of silent AF in a significant number of individuals at risk for stroke compared to routine care (no screening) and will thus lead to improved outcomes through initiation of anticoagulation. The aim of this study is to screen for AF in Native Americans who are seen at the Absentee Shawnee Tribal clinic using a smartphone-based ECG device. Individuals who are at least 50 years old and have no prior history of AF will be eligible for enrollment in the study. Eligible participants will receive a 30-second ECG recording during their visit at the Absentee Shawnee Tribal clinic. The device has an algorithm for diagnosis of AF, which is 98% sensitive and 97% specific. A cardiologist will overread the tracings that are diagnosed by AF by the device. Those confirmed to have AF will be referred to a cardiologist for further evaluation and management. The clinical characteristics of those who are found to have AF will be compared with those who are not, in order to identify risk factors for AF. Newly diagnosed AF using this method is expected to be approximately 2.5%. We aim to include a total of 1,500 participants over 12 months. The proposed study will provide the basis for the design of further intervention studies using mobile technology to improve the health of Native Americans and other minority populations. In light of the high prevalence of risk factors for AF in Native Americans and the association of silent AF with stroke, this novel approach for AF screening has the potential to impact clinical practice and improve health outcomes among a large number of individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50 or older

Exclusion Criteria:

* Known history of atrial fibrillation

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
incidence of newly diagnosed atrial fibrillation | 12 months

SECONDARY OUTCOMES:
prevalence of guideline-directed anticoagulant use among participants who are found to have atrial fibrillation | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stavrakis S, Elkholey K, Lofgren MM, Asad ZUA, Stephens LD, Freedman B. Screening for Atrial Fibrillation in American Indian Adults in a Tribal Primary Care Clinic. J Am Heart Assoc. 2021 May 4;10(9):e020069. doi: 10.1161/JAHA.120.020069. Epub 2021 Apr 21. PMID 33878888